CLINICAL TRIAL: NCT01658020
Title: Clinical Trials to Evaluate Efficacy and Safety of Zabofloxacin Tablet 400mg and Moxifloxacin Tablet 400mg After Multi-dose Oral Administration in Patients With Acute Bacterial Exacerbation of Chronic Obstructive Pulmonary Disease.
Brief Title: A Study to Evaluate Efficacy and Safety Profile of Zabofloxacin Tablet 400mg and Moxifloxacin Tablet 400mg
Acronym: DW224-III-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Collaborators: Chonbuk National University Hospital (Other); Chosun University Hospital (Other); Bundang CHA Hospital (Other); Chungbuk National University (Other); Kangdong Sacred Heart Hospital (Other); Hanyang University (Other); Asan Medical Center (Other); Gachon University Gil Medical Center (Other); The Catholic University of Korea (Other); Konyang University Hospital (Other); KangWon National University Hospital (Other); Gyeongsang National University Hospital (Other); Kyunghee University Medical Center (Other); Korea University Anam Hospital (Other); DongGuk University (Other); Severance Hospital (Other); Yeungnam University Hospital (Other); Ulsan University Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Inje University (Other); Chonnam National University Hospital (Other); Catholic University of Korea Saint Paul's Hospital (Other); Incheon St.Mary's Hospital (Other); Masan Samsung Hospital, South Korea (Other); Konkuk University Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Wonju Severance Christian Hospital (Other); Hallym University Medical Center (Other); Ajou University (Other); Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW224-III-3
Record Dates: First submitted 2012-07-25; First posted 2012-08-06 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute exacerbation of Chronic obstructive pulmonary disease; Acute Exacerbation; Chronic obstructive pulmonary disease(COPD); Zabofloxacin; Moxifloxacin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — zabofloxacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DW224 (Experimental): Zabofloxacin 367mg tablet P.O. once daily for 5days and then Placebo P.O. once daily for 2days
  Interventions: Drug: Zabofloxacin
- Avelox (Active Comparator): Moxifloxacin 400mg tablet P.O. once daily for 7days
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Zabofloxacin — Zabofloxacin 367mg tablet P.O. once daily for 5days and then Placebo P.O. once daily for 2days
  Other Names: DW224
  Arms: DW224
Drug: Moxifloxacin — Moxifloxacin 400mg tablet P.O. once daily for 7days
  Other Names: Avelox
  Arms: Avelox

SUMMARY:
The purpose of this study is to Evaluate the Efficacy and Safety Profiles of oral multiple dose of Zabofloxacin Tablet 400 mg.

DETAILED DESCRIPTION:
A Phase 3, Multicenter, Double Blind, Active Controlled, Randomized Study to Evaluate the Efficacy and Safety of Zabofloxacin for Patients with acute bacterial exacerbation of Chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female same or older than age of 40
* Severity of acute exacerbation of Chronic obstructive pulmonary disease(COPD) must suit oral administration treatment
* Diagnosed as COPD before receiving written informed consent and outcome measure of spirometry testing confirmed as [Ratio of Forced Expiratory Volume in 1 second(FEV1) to Forced Vital Capacity(FVC)](FEV1/FVC) < 0.7
* Subject showing following signs and symptoms:

  (i)Purulent Sputum or Sputum level is increased (ii)Difficulty in breathing is increased
* Female subjects who might be pregnant must do pregnancy test and results should be negative before randomization is done. She must receive written informed consent form (NOTE: Subject who has used single hormone contraception for pregnancy control or has not been more than 1 year after Tubule ligation and menopause are excluded from the study)
* Subject who can agree and sign written informed consent form approved by Institutional Review Board(IRB) before participating in study and follow study requirements

Exclusion Criteria:

* Subject who administered excess daily dose of antimicrobial/antibiotics in past 72 hours before receiving written consent
* Diagnosed to have pneumonia by taking chest X-ray in past 48 hours before receiving written consent
* Diagnosed to have infectious diseases or such diseases results in complications before receiving written consent (NOTE: Septic shock, Bronchiectasis, Lung abscess, Pneumonia, Active tuberculosis, Pulmonary malignancy, Cystic fibrosis, Empyema, Asthma)
* Have kidney or liver diseases who correspond following criteria:

  (i) Creatinine Clearance(CCr) < 50 mL/min (ii) Blood Urea Nitrogen(BUN) ≥ 30 mg/dl (iii) Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 3 x Upper Limit Normal(ULN) (iv) Total bilirubin > 2 x ULN (v) Alkaline Phosphatase(ALP) > 2 x ULN.
* Organic gastrointestinal disorder having abnormal absorption problem condition in past 6 months before receiving written consent (NOTE: Active Crohn's disease, active ulcerative colitis)
* Diagnosed to have neutropenia where absolute neutrophil count is < 1,000cells/mm3 (NOTE: Even though subject neutrophil count is < 1,000cells/mm3, if it is acute infection, subject maybe possible to participate)
* Chronic Hepatitis B carrier
* Have proof that subject is Hepatitis C carrier or have Hepatitis C antibody
* Immunodeficiency diseases such as HIV positive, AIDS, Bone marrow transplant or leukemia
* Have medical history of hypersensitive reaction to antibiotics of fluoroquinolones
* Have medical history of seizure or administration of anti-seizure drug in past 1 year before receiving written consent (NOTE: Epilepsy, Convulsions, Myasthenia gravis)
* Medical history of ventricular arrhythmia
* Medical history of QTc prolongation or currently administering drug that delays QTc interval (NOTE: QTc prolongation means QTc interval > 450 msec)
* Complex infections or diseases that can effect study assessment or need long-term antibiotic treatment exceeding 7 days
* Subject who has participated in Clinical trials or Bioequivalence test in past 30 days before receiving written consent
* Clinically significant by observations considered as unsuitable based on medical judgement by investigators where current condition can effect quality of safety or data

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeon-Mok Oh, M.D., Principal Investigator — Asan Medical Center; Sang-Do Lee, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yoon S, Kim TE, Kim TH, Na JO, Shin KC, Rhee CK, Jung SS, Choe KH, Yoo KH. Clinical Role of the Chronic Obstructive Pulmonary Disease Assessment Test in Prediction of the Response to Treatment for Exacerbations. J Korean Med Sci. 2020 Jan 13;35(2):e10. doi: 10.3346/jkms.2020.35.e10. PMID 31920016
- See also: Asan Medical Center — http://medical.amc.seoul.kr/medservice/main/main.do
- See also: Dong Wha Pharm. Co. Ltd. — http://www.dong-wha.co.kr/dw_main.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- DW224: Zabofloxacin 400mg tablet P.O. once daily for 5days and Placebo P.O. once daily
Period: Overall Study
Arm/Group | DW224 | Avelox
Started | 175 | 167
Completed | 167 | 158
Not Completed | 8 | 9
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- DW224: Zabofloxacin 367mg tablet P.O. once daily for 3 days and then placebo P.O. once daily for 2 days
- Avelox: Moxifloxacin 400mg tablet P.O. once daily for 7 days
- Total: Total of all reporting groups
Arm/Group | DW224 | Avelox | Total
Number analyzed (Participants) | 175 | 167 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.76 (7.79) | 68.40 (8.04) | 68.07 (7.91)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 93 | 190
  >=65 years | 78 | 74 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 8 | 30
  Male | 153 | 159 | 312
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 175 | 167 | 342

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response in the Clinical Populations
Description: Clinical response corresponding clinical cure at Test of Cure visit. Based on the clinical outcomes, the results of assessment were classified into Clinical Cure, Clinical Failure, Relapse and Indeterminate.
Time Frame: 10days
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DW224: Zabofloxacin 367mg tablet P.O. once daily for 5 days and then placebo P.O. once daily for 2 days
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 143 | 131
percentage of participants | 86.71 [81.15 to 92.28] | 86.26 [80.36 to 92.16]

2. Secondary Outcome: Clinical Response in the Clinical Population
Description: Clinical response corresponding clinical cure at End of Study visit. Based on the clinical outcomes, the results of assessment were classified into Clinical Cure, Clinical Failure, Relapse and Indeterminate.
Time Frame: 36days
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Avelox: Moxifloxacin 400mg tablet P.O. once daily 7 days
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 143 | 131
percentage of participants | 76.22 [69.25 to 83.20] | 70.99 [63.22 to 78.76]

3. Secondary Outcome: Clinical Cure Rate in the Microbiological Per Protocol(PP) Population
Description: Clinical response corresponding clinical cure in the microbiological per-protocol population.
  Microbiological responses were discriminated for the pathogens isolated from the respiratory secretion samples of subjects.
Time Frame: 10days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 43 | 39
Percentage of participants | 88.37 [78.79 to 97.95] | 94.87 [87.95 to 100.00]

4. Secondary Outcome: Microbiological Response Rate
Description: Microbiological response rate in the microbiological per protocol(PP) population.
  Microbiological rate were discriminated for the pathogens isolated from the respiratory secretion samples of subjects.
Time Frame: 10days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 43 | 39
Percentage of participants | 67.44 [53.44 to 81.45] | 79.49 [66.81 to 92.16]

5. Secondary Outcome: Change in EXACT-PRO Score
Description: The outcome measurement is Change in EXACT-PRO score for clinical populations at Test of cure visit.
  EXACT-PRO means that the questionnaires for Exacerbation of Chronic Pulmonary Disease Tool-Patient Reported Outcome of United BioSource Corporation(UBC) of USA that had been standardized, equipped with reliability and feasibility applicable to various COPD patients groups were used in order to quantitate frequency, severity and duration of acute exacerbation as a tool to measure acute exacerbation of COPD.
  EXACT-PRO is consisted of 14 questionnaire items were classified into 3 domains, Respiratory Distress Domain, Cough/Sputum Domain, and Chest Symptoms Domain. The Scores of each domain were to be summed into the domain raw summed score or converted into EXACT domain score according to the conversion table. The total score had value in the range from 0 to 100 and higher the value was, severer the respiratory symptoms were in evaluation.
Time Frame: 10 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 141 | 130
scores on a scale | -6.90 (9.59) | -4.29 (9.72)

6. Secondary Outcome: Change in CAT Scores
Description: The outcome measurement is Change in CAT scores for clinical populations at Test of cure visit.
  CAT score means that COPD Assessment Test was used as a tool to assess the effects of COPD on physical, mental status and daily life.
  CAT is consisted of 8 items in total and each question item was scored from 0 point to 5 point.
  The scores of each question item were summed into the total score, which had values between 0 and 40.
Time Frame: 10 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | DW224 | Avelox
Number analyzed (Participants) | 139 | 130
scores on a scale | -4.46 (5.88) | -2.48 (5.96)

ADVERSE EVENTS:
Time Frame: About 1.5 years
Groups:
- DW224: Zabofloxacin Tablet 400mg given by oral administration
  Moxifloxacin Tablet 400mg: multiple-dose
- Avelox: Moxifloxacin Tablet 400mg given by oral administration
  Zabofloxacin Tablet 400mg: multiple-dose
Arm/Group | DW224 | Avelox
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/167
Other Adverse Events (participants affected / at risk) | 17/175 | 16/167
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DW224 (N=175) | Avelox (N=167)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vimiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Red blood cell microcytes present (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less